CLINICAL TRIAL: NCT02697968
Title: Electroacupuncture for Relieving Pain in Ankylosing Spondylitis: a Single-arm Pilot Study
Brief Title: Electroacupuncture for Relieving Pain in Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor LAO Lixing, Director, School of Chinese Medicine, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 15-458
Record Dates: First submitted 2016-02-24; First posted 2016-03-03 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Electroacupuncture

ARMS (1):
- Electroacupuncture (Experimental)
  Interventions: Device: Electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture

SUMMARY:
Background: Ankylosing spondylitis imposes burdens on individuals and society that AS costs 3 times higher than general population. Conventional approaches for AS have their limitation. Previous studies demonstrated acupuncture has significant therapeutic effects for AS in diminishing joint pain, enhancing functional disorders and modifying spinal deformity. Although acupuncture is effective in relieving pain in AS patients, the evidence is very limited due to methodological flaws.

Design This study will be a single-arm pilot study in patients with AS. Eligible subjects will receive electroacupuncture treatment twice per week for at least 6 weeks (12 sessions in total). The length of treatment can be extended to a maximum of 10 weeks (20 sessions in total) if participants request a prolonged treatment. The acupuncturist, who is a registered Chinese medicine practitioner, of this trial will not participate in data collection and data entry.

Objective: To explore the treatment effect of electroacupuncture for relieving pain in ankylosing spondylitis.

Setting: Hong Kong

Participants: 20 subjects with a diagnosis of ankylosing spondylitis

Main Measures: Pain Severity Numerical Rating Scale (NRS), Adverse events

Data analysis All data will be double-entered and checked for consistency before conducting the analysis. Binomial test will be used to analyze the percentage of responders to treatment compared with a reference value of 10%. Wilcoxon signed rank test will be used to compare the values of all continuous variables between baseline and post treatment. The population for safety analyses will include all subjects who receive at least one acupuncture treatment. Adverse events will be coded using the WHO Adverse Reaction Terminology Dictionary. Special attention will be given to those subjects who have discontinued treatment due to adverse events or who experience serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. with a diagnosis of AS and fulfilled either ASAS criteria or Modified New York criteria,
2. Bath Ankylosing Spondylitis Disease Activity Index, BASDAI ≥4,
3. currently taking analgesic or NSAIDs for pain control,
4. spinal pain assessment score≥4 on a numerical rating scale (NRS; 0-10 scale)

Exclusion Criteria:

1. having active skin lesion or open wound over the needle placement areas;
2. having heart disease, bleeding disorder or taking anticoagulant drugs
3. have previous acupuncture experience 12 months before the baseline,
4. are pregnant, breast-feeding or of childbearing potential but not using adequate contraception;
5. having psoriasis, rheumatoid arthritis, osteoarthritis, psoriatic arthritis or reactive arthritis;
6. having unstable medical condition such as liver and/or kidney failure or cancers.;
7. concurrently taking or injecting steroid.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Pain Severity Numerical Rating Scale (NRS) | week 0 and 6

SECONDARY OUTCOMES:
Types and dosage of drug(s) intake | week 0, 2, 4, 6, 8, 10, 12, 14 and 18
Bath Ankylosing Spondylitis Functional Index (BASFI) | week 0, 6, 10 and 18
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | week 0, 6, 10 and 18
Bath Ankylosing Spondylitis Global Index (BASGI) | week 0, 6, 10 and 18
Quality of life of patients as evaluated by SF-36 | week 0, 6, 10 and 18
  Quality of life of patients will be measured.
Bath Ankylosing spondylitis Metrology Index (BASMI) | week 0, 6, 10 and 18
Chest expansion as measured by the change in circumference at 4th intercostal level between maximal inspiration and expiration in cm | week 0, 6, 10 and 18
Joints count | week 0, 6, 10 and 18
C-reactive protein (CRP) | week 0, 6, 10 and 18
Erythrocyte sedimentation rate (ESR) | week 0, 6, 10 and 18
Change in Pain Severity Numerical Rating Scale (NRS) | week 0, 2, 4, 8, 10, 12, 14, and 18

OTHER OUTCOMES:
Number of patients withdraw and the corresponding reasons | 18 weeks
Number of subjects with and corresponding types of adverse events | 18 weeks
Treatment Credibility by the Credibility of Treatment Rating Scale (CTRS) | Week 0,6 and 10

CONTACTS AND LOCATIONS:
Overall Officials: Lixing LAO, Ph.D., Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong